CLINICAL TRIAL: NCT02859077
Title: EGFR-TKI With Chemotherapy as First Line Treatment in Stage IIIB/IV NSCLC Patients With Both EGFR Mutation and BIM Deletion Polymorphism
Brief Title: EGFR-TKI With Chemotherapy in NSCLC Patients With Both EGFR Mutation and BIM Deletion Polymorphism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Prof. Caicun Zhou, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPH01
Record Dates: First submitted 2016-07-31; First posted 2016-08-08 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: NSCLC; BIM; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Gemcitabine; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGFR-TKI and Chemotherapy (Experimental): NSCLC patients
  Interventions: Drug: EGFR-TKI; Drug: Chemotherapy（pemetrexed/gemcitabine）; Drug: Chemotherapy（carboplatin）

INTERVENTIONS:
Drug: EGFR-TKI — EGFR-TKI (gefitinib)
  Other Names: gefitinib
Drug: Chemotherapy（pemetrexed/gemcitabine） — Chemotherapy (pemetrexed/gemcitabine)
  Other Names: pemetrexed/gemcitabine
Drug: Chemotherapy（carboplatin） — Chemotherapy（carboplatin）
  Other Names: carboplatin

SUMMARY:
BIM deletion polymorphism might be associated with a poor clinical response to EGFR-TKIs in patients who had NSCLC with EGFR mutations. In the study, the investigators want to use EGFR-TKI with chemotherapy as first line treatment in stage IIIB/IV NSCLC patients with both EGFR mutation and BIM deletion polymorphism.

DETAILED DESCRIPTION:
BIM deletion polymorphism was a poor clinical response marker to EGFR-TKIs in NSCLC patients who had EGFR mutations. In the study, the investigators want to use EGFR-TKI with chemotherapy as 1 st treatment in stage IIIB/IV NSCLC patients with both EGFR mutation and BIM deletion polymorphism.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent Age >=18 years Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic Stage IV Non-Small Cell Lung Cancer (NSCLC) A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology) Must have measurable or non-measurable disease Must be able to comply with study and follow-up procedures

Exclusion Criteria:

Small cell, carcinoid, or mixed small cell lung cancer Malignancies within 3 years except for adequately treated carcinoma in situ of -the cervix or basal or squamous cell skin cancer Symptomatic or untreated brain metastases Prior systemic chemotherapy for NSCLC Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or serious cardiac arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible) History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival | 1 year

SECONDARY OUTCOMES:
Overall Response Rate | 1 year
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, PHD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University

IPD SHARING:
Plan to Share IPD: Yes
We will share the analysis data.